CLINICAL TRIAL: NCT05999279
Title: A Cross-sectional Study Addressing Lebanese Patient Preferences With Pharmaceutical Care: Traditional Versus Digital Health?
Brief Title: Patient Preferences With Pharmaceutical Care: In-person Versus Digital Health
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Primary investigator, Lebanese University
Other Study IDs: 12/23/D
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Patient Preference
Keywords: pharmaceutical care; preference; digital care
MeSH Terms: conditions — Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Convenient sampling of patients who took at least one medication in the past month
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Developed questionnaire to assess the literacy of patients + another survey to assess their preferences regarding traditional versus digital pharmaceutical care

SUMMARY:
Digital pharmaceutical care, also known as e-pharmaceutical care or telepharmacy, refers to using digital technologies to provide remote pharmaceutical care services. It involves the application of digital tools and platforms to deliver medication-related services, patient counseling, medication management, and other pharmaceutical care activities. It allows patients to access pharmaceutical services conveniently from their homes or any location with an internet connection. This is particularly beneficial for individuals with limited mobility, those living in rural or underserved areas, or patients with difficulty visiting a physical pharmacy. However, it is essential to note that while digital pharmaceutical care provides many benefits, it may only suit some patients or situations. Some individuals may still prefer face-to-face interactions or may require hands-on assistance, especially for complex medication management. Healthcare providers should assess the appropriateness of digital solutions on a case-by-case basis and ensure patient privacy and data security when implementing digital pharmaceutical care services.

ELIGIBILITY:
Inclusion Criteria:

* Patients who took at least one medication in the past month
* Patient visiting two community pharmacies

Exclusion Criteria:

* Those refusing to participate
* Those with severe hearing or mental problems

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals who visited two community pharmacies during the data collection period. No criteria were based on sex, race, nationality, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Patient preference | through study completion, an average of 2 months
  A self-reported questionnaire was developed and piloted on the first 30 patients visiting the pharmacies. Minor modifications were performed taking into consideration two expert reviews. It is available in Arabic (native language) and English based on participants' preferences. It includes 3 parts: the first part comprises the baseline characteristics of the patients and their medical history/habits; the second part reports patients' preferences, benefits and disadvantages of each of the outcomes (in-person versus digital health); and the third part assess e-literacy among them using the e-HEALS 8-item scale previously validated on the Arab population.

CONTACTS AND LOCATIONS:
Locations (2):
- Lebanon (2):
  - Pharmacy Bouchi, Beirut, Mount Lebanon
  - Pharmacy du Liban, Beirut

IPD SHARING:
Plan to Share IPD: No